CLINICAL TRIAL: NCT01308866
Title: Effectiveness of a Shared Decision Aid Tool for Cardiovascular Risk Prevention in Hypercholesterolemic Patients
Acronym: PLEGATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Preventive Services and Health Promotion Research Network (Other)
Responsible Party: Joan Gene Badia, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PLEGATS
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-03

CONDITIONS: Hypercholesterolemia; Cardiovascular Risk
Keywords: cardiovascular diseases; patient education; primary health care; consumer participation; decision aids
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Usual care
- Intervention (Experimental): Intervention arm using a share-decision tool for cardiovascular patients
  Interventions: Behavioral: Share decision tool

INTERVENTIONS:
Behavioral: Share decision tool
  Arms: Intervention

SUMMARY:
BACKGROUND: Mediterraneans have traditionally a low cardiovascular risk, although emerging lifestyles might change the trend. The aim of this study is to assess if hypercholesterolemic patient involvement in the preventive decision with the help of a decision aid has an impact on cardiovascular (CV) risk reduction superior to usual care.

METHOD: The design is a cluster randomised clinical trial. Participants are hypercholesterolemic patients (>200 mg/dl or c-LDL>130) from four primary care teams of Barcelona. Patients with previous CV events, age over 75 years or cognitive impairment are excluded. It is expected to create two cohorts of 139 patients each one. The randomisation is by doctor. Intervention group will receive information about their CV risk and the risk and benefits of different preventive measures. They will have access to a decission aid that will help them in the choice of the preventive measures.The material (printed and software) is adapted to the Catalan Population using local CV risk tables and will meet the CREDIBLE and DISCERN criteria. STUDY VARIABLES: Sociodemographic variables, CV risk factors, subjective health (SF 12), decisional conflict, anxiety/depression, analytic controls, treatment, treatment adherence, compliance and resources use. Basal evaluation and 3, 6, 12 month assessment. The study, financed by FIS, will begin the 01-07-2007.

RESULTS: The expected results are a higher reduction on the CV risk factors in the intervention group versus regular care.

CONCLUSIONS Study will provide a tool to be used in Spanish and Catalan population.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 14 and 75 years old having the inclusion criteria and consulting for cardiovascular risk diseases (CVD) in these centers.
* Patients who allow to participate in this study

Exclusion Criteria:

* Patients with mental disorders.
* Secundary cardiovascular risk patients

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2007-07; Primary Completion 2010-09 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Cardiovascular risk reduction | one year
  Cardiovascular risk reduction measured throught REGICOR Spanish scale

SECONDARY OUTCOMES:
Life self-perceived quality | one year
  Throught questionnaire SF-12
Anxiety and depression | one year
  Throught HADS scale
Decision empowerment | one year
  Otawa's decision scale

CONTACTS AND LOCATIONS:
Overall Officials: Joan Gene-Badia, MD, PhD, Principal Investigator — University of Barcelona, CAPSE, Health Policy Monitor; Patricia Fernandez-Vandellos, RN, MpH, Study Chair — University of Barcelona
Locations (2):
- Spain (2):
  - Capse-Gesclínic, Barcelona, Barcelona
  - Cap El Castell, Castelldefels